CLINICAL TRIAL: NCT07234669
Title: Dietitian-supported Meal-ordering and Systematic Nutritional Care
Status: Completed | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01
Record Dates: First submitted 2023-05-10; First posted 2025-11-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Diseases; Malnutrition
MeSH Terms: conditions — Lung Diseases; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The study investigates whether clinical dietitians at a hospital ward can improve patients' dietary intake during hospitalisation, and whether it can prevent patients from being admitted efter discharge and improve their prognosis. Dietary intake will be measured daily and readmittance within 30 days from discharge will be registered. Questionnaires will be used to assess patients' satisfaction with nutritional care during hospitalisation.

DETAILED DESCRIPTION:
Clinical dietitians have been an integrated part of the medical pulmonary ward at Gødstrup Hospital since early 2022. They carry out nutritional screening, nutritional treatment and assisst and guide patients in ordering of meals from the hospital's flexible á la carte food service concept.

The study aims to evaluate the effect of the clinical dietitians' effort on patients nutritional intake, risk of readmittance after discharge and 30-days mortality.

The study is observational, and no changes to the current standard of nutritional care will be implemented throughout the study period. Nutritional intake will be measured daily throughout hospitalisation. Readmittances and vital status will be measured at day 30.

To evaluate the effect of the dietitians' effort, data will be compared to historical data from a previous completed study at the same ward.

Patient satisfaction with nutrional care during hospitalisation will be measured with a purpose-designed questionnaire.

Informed written consent will be obtained from all patients before inclusion, and they will be informed that their partitipation is voluntary and that they can withdraw their consent at anytime.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted at the medical pulmonary ward
* Expected admittance of minimum 48 hours
* At nutritional risk defined as a Nutritional Risk Screening 2002 Score of >=3
* Able to understand and speak Danish

Exclusion Criteria:

* Terminal illness
* Dementia
* Enteral or parenteral nutrition
* Need of texture-modified diet or other special diets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at nutritional risk admitted to the pulmonary medical ward at Gødstrup Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Nutritional intake | Through study completion, an average of 5 days
  Mean daily energy and protein intake in percentage of estimated requrements

SECONDARY OUTCOMES:
Length of hospital stay | Through study completion, an average of 5 days
  Number of days from admission date at the pulmonary ward to discharge.
Readmission | Measured at day 30
  Number of participants that have been readmitted after discharge
30-days mortality | Measured at day 30
  Measured as vital status at follow-up
Patients' experience of whether they received nutritional guidance during hospitalisation | Measured at day of discharge, on average day 5
  The degree to which patients experience to have received nutritional guidance measured on 5-point Likert scales (5 indicating very high degree, 1 indicating very low degree)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne B Kristensen, PhD, Principal Investigator — Gødstrup Hospital
Locations (1):
- Gødstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No